CLINICAL TRIAL: NCT05216965
Title: Phase I/II Clinical Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of 9MW2821 in Subjects With Advanced Malignant Solid Tumors
Brief Title: A Clinical Study of 9MW2821 in Subjects With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-2021-CP102
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9MW2821 (Experimental)
  Interventions: Drug: 9MW2821

INTERVENTIONS:
Drug: 9MW2821 — All subjects will receive a single intravenous (IV) infusion of 9MW2821 once weekly for the first 3 weeks of every 4 week cycle (i.e., on Days 1, 8 and 15).

SUMMARY:
This study is a Phase 1/2, first-in-human, open-label, dose-escalation and cohort expansion study designed to characterize the safety, tolerability, pharmacokinetics, preliminary antitumor activity and immunogenicity of 9MW2821 administered by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
2. Male or female subjects aged 18 to 80 years (including 18 and 80 years).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically or cytologically confirmed advanced malignant solid tumors (except sarcoma).
5. For Cohort Expansion: Subjects must submit tumor tissue for Nectin-4 expression.
6. Life expectancy of ≥ 3 months.
7. Subjects must have measurable disease according to RECIST (version 1.1).
8. Adequate organ functions.
9. Sexually active fertile subjects, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.
10. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. Chemotherapy or radiotherapy within 21 days prior to the first dose of study drug, or any other anticancer therapy within 14 days prior to the first dose of study drug.
2. Preexisting treatment related toxicity Grade ≥ 2 (except alopecia).
3. Major surgery within 28 days prior to first dose of study drug.
4. History of uncontrolled diabetes mellitus.
5. Preexisting peripheral neuropathy Grade ≥ 2.
6. Received treatment of nectin-4 targeted ADC with MMAE payload.
7. Any live vaccines within 4 weeks before first dose of study drug or during the study.
8. Documented history of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
9. Other severe or uncontrolled disease, i.e. severe respiratory system disease, thromboembolic events, active bleeding or active infection.
10. Uncontrolled central nervous system metastases.
11. History of another malignancy within 3 years before the first dose of study drug. Subjects with curable malignancies are allowed.
12. History of autoimmune disease requiring systemic treatment within 2 years before the first dose of study drug.
13. Has ocular conditions that may increase the risk of corneal epithelium damage.
14. Known sensitivity to any of the ingredients of the investigational product; History of drug abuse or mental illness.
15. Any P-glycoprotein (P-gp) inducers/inhibitors or CYP3A4 inducers/inhibitors within 14 days prior to the first dose of study drug
16. Use of any investigational drug or device within 2 months prior to the first dose of study drug.
17. Condition or situation which may put the subject at significant risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2022-06-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days post last drug administration
Objective Response Rate (Phase 2) | Up to 24 months
  Defined as the percentage of subjects who experience a best response of either CR or PR. CR and PR must be confirmed ≥ 28 days later.

SECONDARY OUTCOMES:
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Maximum observed concentration (Cmax)
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Area under the concentration-time curve (AUC)
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Half-life (t1/2)
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Clearance (CL)
Disease Control Rate | Up to 24 months
  Defined as the percentage of subjects who experience a best response of CR, PR or stable disease (SD)
Duration of Response | Up to 24 months
  Time from the date of the first complete response (CR) or partial response (PR) to the earliest date of disease progression or death from any cause. DOR is only defined for subjects who have best overall response of CR or PR.
Time to Response | Up to 24 months
  Time from the date of first infusion to the date of confirmed CR or PR
Progression Free Survival | Up to 24 months
  Time from the date of first infusion to the earliest date of documented disease progression per radiological evidence or death from any cause
Overall Survival | Up to 24 months
  Time from the date of first infusion until the date of death from any cause.
Incidence of Anti-Drug Antibody (ADA) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Liu R, Wang S, Feng Z, Yang H, Gao S, Li X, Yao X, Chen J, Gong Z, Li Y, Li X, Wang S, Hu C, Liu J, Zhang M, Yuan F, Shi B, Lou H, Zhao P, Qiu F, Guo H, Hu B, Xu D, Huang H, Zhang X, Feng M, Wang X, Li G, Liu D, Chen X, Wang P. Bulumtatug Fuvedotin (BFv, 9MW2821), a next-generation Nectin-4 targeting antibody-drug conjugate, in patients with advanced solid tumors: a first-in-human, open-label, multicenter, phase I/II study. Ann Oncol. 2025 Aug;36(8):934-943. doi: 10.1016/j.annonc.2025.04.009. Epub 2025 Apr 25. PMID 40288679